CLINICAL TRIAL: NCT00555282
Title: Rate of Catheter Colonization and Risk of Bloodstream Infection During Use of a Standard Central Venous Catheter (CVC) in Comparison to a Coated CVC
Brief Title: Rate of Catheter Colonization and Risk of Bloodstream Infection During Use of Two Different Central Venous Catheters (CVC)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Dr. Ute Brauer, B. Braun Melsungen AG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HC-G-H-0507
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-02

CONDITIONS: Bacteriaemia; Catheter Related Bloodstream Infection
Keywords: central venous catheter; cvc; coated catheter; bacteriaemia; bloodstream infection
MeSH Terms: conditions — Sepsis | interventions — Central Venous Catheters

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): coated central venous catheter
  Interventions: Device: central venous catheter
- 2 (Active Comparator): standard central venous catheter
  Interventions: Device: central venous catheter

INTERVENTIONS:
Device: central venous catheter — coated central venous catheter
  Other Names: Certofix Protect
  Arms: 1
Device: central venous catheter — standard central venous catheter
  Other Names: Certofix Trio
  Arms: 2

SUMMARY:
The use of these catheters is associated with infectious complications that are an important iatrogenic source of morbidity and mortality. Certofix® protect is a catheter with a surface modified in order to reduce colonization by bacteria. This clinical trial is performed to compare the safety and efficacy of the coated central venous catheter, Certofix® protect, with that of the non-coated standard catheter Certofix®.

DETAILED DESCRIPTION:
Central venous catheters are an essential part of patient management in the ICU (Intensive Care Unit). The use of these catheters is associated with infectious complications that are an important iatrogenic source of morbidity and mortality. Many catheters become colonized with bacteria but only a proportion of colonised catheters go on to cause bacteriemia and sepsis. It is currently impossible to prospectively identify which of the catheters will become colonized and lead to sepsis. Various types of antiseptic or antimicrobial vascular catheter coatings have been developed. Studies showed that the coated catheters were effective in limiting the catheter colonization rate and that they may decrease the risk of catheter-related bloodstream infections. The "Certofix protect" was developed by B.Braun to reduce the risk of catheter related infections. It is a catheter with a modified surface that consists of a high molecular weight polymer which is non-covalently linked to the polyurethane catheter material. This clinical trial is performed to compare the safety and efficacy of the coated central venous catheter, Certofix® protect, with that of the non-coated standard catheter Certofix®.

ELIGIBILITY:
Inclusion Criteria:

* Patients with probable ICU stay
* Patient's first or second catheter placement during actual hospital stay
* Anticipated indwelling central venous catheter period >= 3 days (jugular vein, subclavian vein)
* >= 18 years of age
* Written informed consent of patient or independent physician prior to the participation; in this case: written informed consent after recovery if possible

Exclusion Criteria:

* The catheter will not be placed in the femoral vein
* Inflammation of the skin at the site of puncture prior to puncture
* Known hypersensitivity to any of the components (i.e. polyhexanide or related substances such as chlorhexidine)
* Participation in another clinical trial
* Emergency insertion of catheter in the field

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2005-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Incidence of catheter colonization | after catheter removal
Incidence of bloodstream infection | during treatment

SECONDARY OUTCOMES:
Safety of catheter: complications related to the catheter and adverse events in general, clinical therapy, TISS-Score, ICU stay, infection markers | until discharge from ICU
Safety of catheter: central venous catheter variables, time of catheter insertion and removal, kind of colonization | catheter removal

CONTACTS AND LOCATIONS:
Overall Officials: Jan Pachl, Prof. Dr., Principal Investigator — Faculty Hospital Charles University Prague; Pavel Sevcik, Prof. Dr., Principal Investigator — Brno University Hospital
Locations (2):
- Czechia (2):
  - Faculty Hospital Brno, Brno
  - Faculty Hospital Charles University, Prague

REFERENCES:
- [Derived] Krikava I, Kolar M, Garajova B, Balik T, Sevcikova A, Roschke I, Sevcik P. The efficacy of a non-leaching antibacterial central venous catheter - a prospective, randomized, double-blind study. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2020 Jun;164(2):154-160. doi: 10.5507/bp.2019.022. Epub 2019 May 28. PMID 31142873